Statistical Analysis Plan

NCT03856177

03/15/2023

In relation to ERP data, we first aimed to conceptually replicate and extend findings by Foti & Hajcak (2010) by assessing whether the RewP was affected by mood. An independent-samples t-test was conducted between mood manipulation groups (sad vs. neutral) to test whether sad mood could relatively reduce the RewP. The RewP was quantified as a reward-specific ERP component at electrode site FCz and amplitude was measured as the average amplitude within a 200–350ms time window. The electrode site and time window were decided a priori based on previous work utilizing the probabilistic selection task to investigate the RewP (Cavanagh et al., 2019). Data were analyzed using the Jamovi toolkit in R. There was no adjustment for multiple comparisons correction.